CLINICAL TRIAL: NCT03761199
Title: The Influence of Cryostimulation on Selected Mediators of Inflammation and on the Level of Lubrication, Moisture and pH of the Skin of Patients With Atopic Dermatitis (AD)
Brief Title: Assessment of the Impact of Whole Body Cryostimulation on Skin Physiological Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: USPEKrakow
Record Dates: First submitted 2018-11-06; First posted 2018-12-03 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2019-11

CONDITIONS: Quality of Life; Atopic Dermatitis
Keywords: AD patients; whole body cryostimulation
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a group of patients with AD (Experimental): 15 people with clinically diagnosed atopic dermatitis (AD), established on the basis of criteria Hanifin and Rajka
  Interventions: Other: whole body cryostimulation
- control group (Other): 15 healthy persons which will form the control group
  Interventions: Other: whole body cryostimulation

INTERVENTIONS:
Other: whole body cryostimulation — In this research project will be performed 15 treatments in cryogenic chamber (1 once a day, every day, with a break on Saturdays and Sundays). Cryostimulation will be conducted in a cryochamber located in the Małopolska Cryotherapy Centre in Kraków, Poland (Polish: Małopolskie Centrum Krioterapii). The whole body cryostimulation (WBC) exposure will be administered in a special temperature-controlled unit which consists of two rooms (-60° and -120°C). Throughout the session, the participants will be under direct supervision of qualified doctor.

SUMMARY:
The aim of the planned study will be to evaluate the effect of repeated cryostimulation treatments on immunological, morphological, and biochemical indicators of the peripheral blood of patients with atopic dermatitis (AD). The aim of the study will be also to measure the oiling, hydration and pH of the skin of patients with AD after a series of treatments in a cryogenic chamber.

Each participant will complete a Brief Questionnaire on Quality of Life, Life Satisfaction Index, Self Evaluation Questionnare and DERMATOLOGY LIFE QUALITY INDEX (before and after the WBC procedures).

DETAILED DESCRIPTION:
In this research project will be performed 15 treatments in cryogenic chamber (1 once a day, every day, with a break on Saturdays and Sundays). Cryostimulation will be conducted in a cryochamber located in the Małopolska Cryotherapy Centre in Kraków, Poland (Polish: Małopolskie Centrum Krioterapii). The whole body cryostimulation (WBC) exposure will be administered in a special temperature-controlled unit which consists of two rooms (-60° and -120°C). Persons with any contraindications (both with AD and healthy) for whole body cryostimulation will be excluded from the study. Patients with AD in treatment by phototherapy, cyclosporin A, oral corticosteroids, which are topical calcineurin inhibitors such as pimecrolimus and tacrolimus and patients during or after immunotherapy, children and adolescents under 18 years of age, breast-feeding mothers and pregnant, patients with inflammatory diseases, infectious, autoimmune and cancer will be excluded from research.

The participants will be informed about how they should breathe and move in the cryochamber. Entry to the cryochamber will be preceded by a 30s acclimatization period in the vestibule at a temperature of -60° C, after which the subjects will go directly to the proper chamber (-120° C) for three minutes. During the procedure, all participants will be clothed in shorts, wool socks, gloves and hats or headbands for protection from frostbite, as well as wooden clogs. Additionally, participants will wear surgical masks with a layer of gauze over the mouth and nose for protection. Throughout the session, the participants will be under direct supervision of qualified doctor.

ELIGIBILITY:
Inclusion Criteria:

* informed consent for research;
* equal age and above 18 years of age;
* no contraindications to cryostimulation procedures;
* clinically diagnosed atopic dermatitis (people with AD);

Exclusion Criteria:

* lack of informed consent for research
* patients with AD in treatment by phototherapy, cyclosporin A, oral corticosteroids, which are topical calcineurin inhibitors such as pimecrolimus and tacrolimus and patients during or after immunotherapy,
* children and adolescents under 18 years of age,
* breast-feeding mothers and pregnant,
* patients with inflammatory diseases, infectious, autoimmune and cancer

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
examination of moisturizing of the skin of each patient (AD group) | 5 minutes before 1st treatment of WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigating. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of moisturizing of the skin of each patient (control group) | 5 minutes before 1st treatment of WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigating. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of greasing of the skin of each patient (AD group) | 5 minutes before 1st treatment of WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigating. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of greasing of the skin of each patient (control group) | 5 minutes before 1st treatment of WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigating. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of the pH level of the skin of each patient (AD group) | 5 minutes before 1st treatment of WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigating. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of the pH level of the skin of each patient (control group) | 5 minutes before 1st treatment of WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigating. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of moisturizing of the skin of each patient (AD group) | 5 minutes after 15th WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigating. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of moisturizing of the skin of each patient (control group) | 5 minutes after 15th WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigating. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of greasing of the skin of each patient (AD group) | 5 minutes after 15th WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigatinhg. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of greasing of the skin of each patient (control group) | 5 minutes after 15th WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigatinhg. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of pH level of the skin of each patient (AD group) | 5 minutes after 15th WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigating. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of pH level of the skin of each patient (control group) | 5 minutes after 15th WBC
  using special device to the skin test (Courage - Khazaka Electronic, Köln), non-invasive skin tests investigating. Each patient will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of moisturizing of the skin of each patient (AD group) | 3 weeks from completion of treatments in the cryogenic chamber
  using special device to the skin test (Courage - Khazaka Electronic, Köln),non-invasive skin tests investigating. Each subject will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of moisturizing of the skin of each patient (control group) | 3 weeks from completion of treatments in the cryogenic chamber
  using special device to the skin test (Courage - Khazaka Electronic, Köln),non-invasive skin tests investigating. Each subject will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of greasing of the skin of each patient (AD group) | 3 weeks from completion of treatments in the cryogenic chamber
  using special device to the skin test (Courage - Khazaka Electronic, Köln),non-invasive skin tests investigating. Each subject will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of greasing of the skin of each patient (control group) | 3 weeks from completion of treatments in the cryogenic chamber
  using special device to the skin test (Courage - Khazaka Electronic, Köln),non-invasive skin tests investigating. Each subject will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of pH level of the skin of each patient (AD group) | 3 weeks from completion of treatments in the cryogenic chamber
  using special device to the skin test (Courage - Khazaka Electronic, Köln),non-invasive skin tests investigating. Each subject will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.
examination of pH level of the skin of each patient (control group) | 3 weeks from completion of treatments in the cryogenic chamber
  using special device to the skin test (Courage - Khazaka Electronic, Köln),non-invasive skin tests investigating. Each subject will have a measurement on the inside of the forearm. The measuring probes will be applied directly to the skin. The result will be read on the measuring device.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Kępińska, PhD, Principal Investigator — University of Physical Education in Krakow, Poland; Anna Misiorek, PhD, Principal Investigator — University of Physical Education in Krakow, Poland
Locations (1):
- Magdalena Kępińska, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No